CLINICAL TRIAL: NCT00448331
Title: Facilitated Referral for Children Screening Positive for Mental Illness in the Pediatric Emergency Department and Readiness to Seek Care
Brief Title: Facilitated Referral for Children Screening Positive for Mental Illness
Acronym: MI
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Other Study IDs: 02-9-27; MH063916-03
Record Dates: First submitted 2007-03-14; First posted 2007-03-16 (Estimated); Last update posted 2007-11-02 (Estimated); Status verified 2007-10

CONDITIONS: Mental Disorders; Mentally Ill Persons; Emergency Medicine
Keywords: Mental Disorders; Mentally Ill Persons; Emergency Medicine; Emergency Department; Screening
MeSH Terms: conditions — Mental Disorders; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- positive screen, negative screen: Positive screens are those who received positive feedback regarding their answers to a mental illness screening assessment. Negative screens received feedback stating that they did not screen positive for any mental illness.

SUMMARY:
The purpose of this study is to find out how prevalent unidentified Mental Health issues are in the pediatric population that visits the Emergency Department in an urban city.

DETAILED DESCRIPTION:
The purpose of this research study is to find out how many children in the Emergency Room have emotional issues and how many of them go unnoticed. In particular the study looks at how well a questionnaire for children and teenagers, the DISC Predictive Scales, Version IV (DPS-IV) works and what is the best way to ask the questions. In addition, for children aged 9-17 this study will look at families' readiness to seek care when a problem is indicated.

ELIGIBILITY:
Inclusion Criteria:

* Child Must be With Biological Mother
* Child Presenting to Emergency Department with an Urgent But Stable condition
* Child must be between the ages of 6 years and 18 years
* Child must have no prior history of Behavioral Health concerns or diagnoses

Exclusion Criteria:

* Child has prior Behavioral Health history, diagnosis, or concerns
* Child not between ages of 6 years and 18 years of ages
* Child presenting without Biological Mother present
* Child acuity level outside of Urgent But Stable for presenting complaints

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Emergency Department patients ages 6-18 who present without any history of mental health issues.
Sampling Method: Non-Probability Sample
Enrollment: 551 (Actual)
Dates: Start 2004-06; Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jackie Grupp-Phelan, MD, MPH, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center Emergency Department, Cincinnati, Ohio, United States